CLINICAL TRIAL: NCT07400575
Title: Multicenter, Retrospective, Real World Study of Anlotinib in Cross-line Treatment of NSCLC and SCLC
Brief Title: Anlotinib in Cross-line Treatment of NSCLC and SCLC
Acronym: NSCLC SCLC
Status: Not yet recruiting | Type: Observational
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Qiming Wang, chief physician, Henan Cancer Hospital
Other Study IDs: 2025-631
Record Dates: First submitted 2026-01-27; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: NSCLC (Advanced Non-small Cell Lung Cancer); SCLC, Extensive Stage
Keywords: Anlotinib; mNSCLC; ES-SCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- treatment group: Using Anlotinib in Cross-line Treatment of NSCLC and SCLC
- control group: Using Anlotinib in front-line treatment, but using an Anlotinib-free standard regimen in late-line treatment of NSCLC and SCLC

SUMMARY:
Previous studies on bevacizumab in colorectal and ovarian cancers have demonstrated that continued anti-angiogenic therapy after disease progression can still provide clinical benefits. As a typical multi-targeted anti-angiogenic tyrosine kinase inhibitor, anlotinib hydrochloride has been approved in China for second-line or later treatment of advanced soft tissue sarcoma, where it has also shown significant potential. Retrospective studies have indicated the effectiveness of anlotinib in cross-line treatment for sarcoma. However, there is a lack of multi-center real-world studies evaluating the clinical efficacy of anlotinib in cross-line treatment for driver gene-negative advanced metastatic non-small cell lung cancer and extensive-stage small cell lung cancer.

This study aims to evaluate, through a retrospective multi-center study, the efficacy and safety of anlotinib monotherapy or combination regimens in the later-line treatment of driver gene-negative advanced metastatic non-small cell lung cancer and extensive-stage small cell lung cancer after anlotinib treatment failure, providing clinical evidence for cross-line therapy.

ELIGIBILITY:
Inclusion Criteria:

From October 1, 2018 to April 30, 2025, patients meeting all the following criteria will be included in this study:

* Patients must be diagnosed with advanced metastatic non-small cell lung cancer (including squamous cell carcinoma, adenocarcinoma, etc.) or extensive-stage small cell lung cancer during the period from October 1, 2018 to April 30, 2025.
* Patients clinically documented as having driver gene-negative advanced metastatic non-small cell lung cancer or extensive-stage small cell lung cancer, who were treated with anlotinib during the treatment period and continued using anlotinib after disease progression (with at least 4 months of continuous medication records in the medical records), or other immune or chemotherapy drugs.
* Patients who underwent at least one imaging examination within 90 days before reapplication of anlotinib or other immune or chemotherapy drugs after progression during anlotinib treatment, and subsequently had at least two imaging examinations.

Exclusion Criteria:

From October 1, 2018 to April 30, 2025, patients meeting any of the following criteria will be excluded from this study:

* Patients who received other TKI-class anti-angiogenic drugs (including but not limited to bevacizumab, recombinant human endostatin, pazopanib, regorafenib, cabozantinib, sunitinib, sorafenib, apatinib, axitinib, lenvatinib, fruquintinib, vandetanib, cediranib, nintedanib, pralsetinib, selpercatinib, alectinib, ponatinib) before the first application of anlotinib treatment.
* Patients who received other anti-angiogenic drugs (including but not limited to bevacizumab, recombinant human endostatin, pazopanib, regorafenib, cabozantinib, sunitinib, sorafenib, apatinib, axitinib, lenvatinib, fruquintinib, vandetanib, cediranib, nintedanib, pralsetinib, selpercatinib, alectinib, ponatinib) after progression.
* Patients who underwent surgical treatment during anlotinib therapy. - Patients with driver gene positivity.
* Patients with concurrent other malignant tumors. - Pathological subtypes: advanced metastatic non-small cell lung cancer, including but not limited to large cell carcinoma, adenosquamous carcinoma, carcinoid, pulmonary sarcomatoid carcinoma; extensive-stage small cell lung cancer, including but not limited to oat cell type, mixed type, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of patients with advanced metastatic non-small cell lung cancer and extensive-stage small cell lung cancer who were driver gene-negative and had disease progression after anlotinib treatment.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | From first dose date of Anlotinib until the date of progression based on imaging assessment or date of death from any cause, whichever came first, assessed up to 84 months

IPD SHARING:
Plan to Share IPD: No